CLINICAL TRIAL: NCT05716074
Title: The Effect of Low-İntensity Combined Exercises on Fatigue, Balance and Quality of Life in Patients With Early Stage ALS
Brief Title: The Effect of Low-İntensity Combined Exercises in Patients With Early Stage ALS.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Xhennet Muriqi, Researcher, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-74555795-050.01.04-531483
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; balance; fatigue; quality of life
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised-exercise group (Experimental): This group will be given combined low-intensity exercises under the supervision of a physiotherapist.
  Interventions: Other: Supervised exercise
- Home-exercise group (Experimental): This group will exercise at home without the supervision of a physiotherapist.
  Interventions: Other: Home exercise

INTERVENTIONS:
Other: Supervised exercise — The supervised group will be given 10 minutes of warm-up, 10 minutes of breathing exercises, 20 minutes of low endurance combined exercises (stretching, strengthening, strength exercises), 10 minutes of balance and walking training, and 10 minutes of cool-down exercises. Exercise will be applied for 1 hour a day, 3 days a week for 6 weeks.
  Arms: Supervised-exercise group
Other: Home exercise — The home group will be given 10 minutes of warm-up, 10 minutes of breathing exercises, 20 minutes of low endurance combined exercises (stretching, strengthening, strength exercises), 10 minutes of balance and walking training, and 10 minutes of cool-down exercises. Exercise will be applied for 1 hour a day, 3 days a week for 6 weeks in the home.
  Arms: Home-exercise group

SUMMARY:
The aim of this study is to investigate the effects of low-intensity combined exercises on balance, fatigue and quality of life applied to patients with ALS.

DETAILED DESCRIPTION:
Balance problems and signs of fatigue are seen in early-stage ALS patients. While balance problems lead to falls in ALS patients, fatigue also affects a part of their lives. Studies investigating the effects of low-intensity exercise on fatigue, balance, and quality of life in patients with early-stage ALS are rare. This study will investigate the effects of low-intensity combined exercises on balance, fatigue and quality of life in patients with ALS.

Participants will be randomly divided into Supervised and Home groups. Low-intensity exercises will be applied to the home exercise group as a home program for 1 hour a day, 3 days a week, for 6 weeks. Low-intensity exercises will be applied to the supervised exercise group for 1 hour a day, 3 days a week for 6 weeks, accompanied by a physiotherapist. Evaluations will be made at the beginning and at the end of the treatment.

Berg Balance Scale, Fatigue Severity Scale (FSS), Amyotrophic Lateral Sclerosis Assessment Questionnaire-40 (ALSAQ-40) and revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R) will be used to evaluate patients before and 6 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with early-stage ALS by a neurologist
* Disease duration in the range of 1-18 months
* ALSFRS-R score > 24 higher
* Without infectious disease
* Saturation >95
* Heart rate <92

Exclusion Criteria:

* History of other neurological disease
* Inability to walk
* With mechanical ventilation
* People with Heart and Respiratory Insufficiency
* People with neuropsychological or cognitive impairment
* Dyspnea after ALS

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The fatigue severity scale (FSS) | Baseline, (one week before intervention)
  FSS is a self-report scale of nine items examining motivation, physical function, responsibilities, work, family or social life, exercise, fatigue, frequency of problems, and priority of symptoms.
The fatigue severity scale (FSS) | Post-intervention (7th week)
  FSS is a self-report scale of nine items examining motivation, physical function, responsibilities, work, family or social life, exercise, fatigue, frequency of problems, and priority of symptoms.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | Baseline, (one week before intervention)
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks.
Berg Balance Scale (BBS) | Post-intervention (7th week)
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks.
Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40) | Baseline, (one week before intervention)
  The ALSAQ-40 provides scores for 5 scales: physical mobility, activities of daily living and independence, eating and drinking, communication, and emotional reactions.
Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40) | Post-intervention (7th week)
  The ALSAQ-40 provides scores for 5 scales: physical mobility, activities of daily living and independence, eating and drinking, communication, and emotional reactions.
ALS Functional Rating Scale Revised (ALSFRS-R) | Baseline, (one week before intervention)
  ALSFRS-R measures activities of daily living (ADL) and global function for patients with Amyotrophic Lateral Sclerosis.
ALS Functional Rating Scale Revised (ALSFRS-R) | Post-intervention (7th week)
  ALSFRS-R measures activities of daily living (ADL) and global function for patients with Amyotrophic Lateral Sclerosis.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Ela Tarakci, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakirkoy, Turkey (Türkiye)